CLINICAL TRIAL: NCT02441413
Title: Transplant Optimization Using Functional Imaging (TROFI)
Acronym: TROFI_BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLUI-2014-103_BE
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2016-02

CONDITIONS: Bronchiolitis Obliterans; Lung Transplant Rejection
Keywords: HRCT; High Resolution Computed Tomography scans; Functional Respiratory Imaging; FRI; Computed Tomography; CT; Bronchiolitis Obliterans Syndrome; BOS; Lung Transplant
MeSH Terms: conditions — Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HRCT scans (Experimental): HRCT scan will be taken
  Interventions: Radiation: High Resolution Computed Tomography scans

INTERVENTIONS:
Radiation: High Resolution Computed Tomography scans — A HRCT scan at Functional Residual Capacity (FRC) and Total Lung Capacity (TLC) will be taken on visit 1, visit 2, visit 3, visit 4 and visit 5.
  An Upper Airway (UA) scan will be taken on visit 1.
  Other Names: HRCT scan

SUMMARY:
The objective of this study is to detect Bronchiolitis Obliterans Syndrome (BOS) in an early stage using the outcome parameters generated by Functional Respiratory Imaging (FRI). Robust and automated segmentation algorithms will be developed for these parameters, focusing on quantitative computed tomography (CT) image analyses to provide the physician a more sensitive diagnostics tool. The evolution of BOS over time will be monitored using nmon-rigid image registration methods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ 18 years old
* Written informed consent obtained
* Patient who had undergone a lung transplant a year ago or more
* Female patient of childbearing potential who confirm that a contraception method was used at least 14 days before screening visit and will continue to use a contraception method during the study
* The patient must be able to perform the lung monitoring at home
* Patients diagnosed with BOS 0, BOS 0-p or BOS 1

Exclusion Criteria:

* Pregnant or lactating female
* Known history of or active airways or anastomotic complications requiring intervention such as stenting or dilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11-08 (Actual); Study Completion 2016-11-08 (Actual)

PRIMARY OUTCOMES:
Airway Volume (iVaw) using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.
Airway Resistance (iRaw) using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.
Specific Airway Volume (siVaw) using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.
Specific Airway Resistance (siRaw) using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.
Lobe Volumes (iVlobes) using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.
Air Trapping using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.
Internal Lobar Airflow Distribution using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.
Low attenuation or Emphysema Score using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.
Blood Vessel Density or Fibrosis Score using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.
Airway Wall Thickness using FRI | 12 months
  Exploratory imaging endpoints: HRCT scan will be taken at visit 1- visit 5.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, M.D., M.S., Principal Investigator — University Hospital of Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium